CLINICAL TRIAL: NCT05841082
Title: Coronary RevascUlarIzation in Patients With End-StagE Renal Disease on Dialysis in China-Retrospective Registry
Brief Title: Coronary Revascularization in Patients On Dialysis in China-Retrospective Registry
Acronym: CRUISE-R
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Aerospace Center Hospital (Other); Beijing Chao Yang Hospital (Other); Cangzhou Central Hospital of Tianjin Medical University (Unknown); Civil Aviation General Hospital (Other); Dongguan Tungwah Hospital (Other); Emergency General Hospital (Other); Fifth Affiliated Hospital of Xinjiang Medical University (Other); First Central Hospital of Tianjin (Unknown); Fuwai Yunnan Cardiovascular Hospital (Other); Guangdong Provincial People's Hospital (Other); Henan Provincial Chest Hospital (Other); Ningbo No. 1 Hospital (Other); Peking University People's Hospital (Other); Peking University Shougang Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Tianjin Medical University Second Hospital (Other); Shaoxing People's Hospital (Other); Shengjing Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); the First Affiliated Hospital, Harbin Medical University (Unknown); Zhejiang University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); The Third People's Hospital of Chengdu (Other); Tianjin Medical University General Hospital (Other); Tianjin Union Medicine Center (Unknown); Tongji Hospital (Other); West China Hospital (Other); Xuanwu Hospital, Beijing (Other); Wuhan University (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Head of Cardiology, China-Japan Friendship Hospital
Other Study IDs: CRUISE-2020-12-28
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease; End Stage Renal Disease; Dialysis
Keywords: coronary artery disease; end-stage renal disease; cardiac catheterizations; percutaneous coronary intervention; coronary artery bypass grafting; prognosis; metabolic Syndrome; revascularization; optimal medical therapy
MeSH Terms: conditions — Coronary Artery Disease; Kidney Failure, Chronic; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAD: The investigators recruited all consecutive end-stage renal disease patients requiring dialysis who had significant coronary artery disease, defined as 50% or greater stenosis in any of three main coronary arteries or left main coronary artery on visual assessment of the coronary angiogram

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death in end-stage renal disease (ESRD) patients requiring dialysis. There are limited data on clinical characteristics, treatment strategies and outcomes in this special patient population in China. As a nationwide, observational, multicenter cohort study, this study consecutively included ESRD patients on dialysis with significant CAD at 30 tertiary care centers in 12 provinces in China from January 2015 to June 2021. Patient data collected included demographics, comorbidities, cardiac history, cardiac function, location and severity of CAD, procedural information, medications, and clinical events.

ELIGIBILITY:
Inclusion Criteria:

* 50% or greater stenosis in any of three main coronary arteries or left main coronary artery on visual assessment of the coronary angiogram
* Receive peritoneal dialysis or hemodialysis for more than 3 months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study will be selected from January 2015 to June 2021 among 30 tertiary medical centers across 12 provinces in China
Sampling Method: Non-Probability Sample
Enrollment: 1249 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 12-month follow-up
  All-cause deaths include cardiovascular death and non-cardiovascular death. Cardiovascular death is defined as death due to acute myocardial infarction, heart failure, sudden cardiac death, stroke, cardiovascular procedure, or cardiovascular hemorrhage. Non-cardiovascular death: any death not covered by the above definitions, such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide, or trauma.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | From the hospital admission to 12-month follow-up
  A composite of cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke.
Major or clinically relevant nonmajor bleeding | From the hospital admission to 12-month follow-up
  A bleeding event meeting Bleeding Academic Research Consortium criteria type 2, 3, or 5.
Cardiovascular death | From the hospital admission to 12-month follow-up
  Cardiovascular death is defined as death due to acute myocardial infarction, heart failure, sudden cardiac death, stroke, cardiovascular procedure, or cardiovascular hemorrhage.
Non-fatal myocardial infarction | From the hospital admission to 12-month follow-up
  Non-fatal myocardial infarction is confirmed in patients with ischemic symptoms, elevated serum cardiac biomarkers and/or distinctive ECG changes.
Non-fatal myocardial stroke | From the hospital admission to 12-month follow-up
  Non-fatal myocardial stroke is confirmed as a new neurological deficit attributed to a vascular cause in the central nervous system with imaging evidence by computed tomography or magnetic resonance imaging.
Major bleeding | From the hospital admission to 12-month follow-up
  A bleeding event meeting Bleeding Academic Research Consortium criteria type 3, or 5.
Clinically relevant nonmajor bleeding | From the hospital admission to 12-month follow-up
  A bleeding event meeting Bleeding Academic Research Consortium criteria type 2.
Follow-up major adverse cardiovascular and clinical events | From the hospital admission, and up to 10 years
  We will follow up the patients by telephone and outpatient service to know the all-cause mortality (cardiovascular and non-cardiovascular) and cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Jingang Zheng, MD, PhD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie E, Wu Y, Ye Z, He Y, Zeng H, Luo J, Chen M, Pang W, Xu Y, Gao C, Guo X, Cai L, Ji Q, Yang Y, Wu D, Yuan Y, Wan J, Ma Y, Zhang J, Du Z, Yang Q, Cheng J, Ding C, Ma X, Yin C, Fan Z, Tang Q, Li Y, Sun L, Lu C, Chi J, Yao Z, Gao Y, Yu C, Ren J, Zheng J. Percutaneous coronary intervention vs . medical therapy in patients on dialysis with coronary artery disease in China. Chin Med J (Engl). 2025 Feb 5;138(3):301-310. doi: 10.1097/CM9.0000000000003295. Epub 2024 Sep 25. PMID 39317971